CLINICAL TRIAL: NCT05030246
Title: A Phase Ⅱ, Single-arm Study to Evaluate the Efficacy and Safety of Surufatinib Combined With Toripalimab in Peritoneal Metastatic Carcinoma of Gastrointestinal or Primary Peritoneal Cancer
Brief Title: Trial of Surufatinib Combined With Toripalimab in the Treatment of Peritoneal Metastatic Carcinoma of Gastrointestinal or Primary Peritoneal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-012-CH04 IIT-GI
Record Dates: First submitted 2021-08-24; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-07

CONDITIONS: Refractory Metastatic Digestive System Carcinoma; Primary Peritoneal Cancer
MeSH Terms: interventions — surufatinib; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib 250mg/Toripalimab 240mg (Experimental): Surufatinib at a dose of 250mg Qd, with humanized anti-PD-1 monoclonal antibody（Toripalimab） injected intravenously 240mg per 3 weeks until disease progresses or unacceptable tolerability occurs.
  Interventions: Drug: Surufatinib/Toripalimab

INTERVENTIONS:
Drug: Surufatinib/Toripalimab — Surufatinib 250mg will be taken orally once daily continuously through a 21-day cycle of study treatment. Toripalimab 240mg will be intravenously administered on Day 1 of each cycle.
  Other Names: HMPL-012/JS001

SUMMARY:
This is a phase II, single arm, open-label, single-center study to evaluate the efficacy and safety of Surufatinib combined with Toripalimab in patients with peritoneal metastatic carcinoma of gastrointestinal or primary peritoneal cancer.

DETAILED DESCRIPTION:
The study population is about 72 patients with advanced peritoneal metastatic carcinoma of gastrointestinal or primary peritoneal cancer, who fails or cannot tolerate standard therapies. Surufatinib 250 mg once a day (QD) will be orally administrated and Toripalimab 240mg will be intravenously administered every 3 weeks up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent. For Toripalimab, the upper time limit for treatment is 2 years. The primary objective is overall survival (OS) of Surufatinib combined with Toripalimab in patients with advanced solid advanced peritoneal metastatic carcinoma of gastrointestinal or primary peritoneal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced peritoneal metastatic carcinoma of gastrointestinal or primary peritoneal cancer
2. Failed after standard treatment
3. Have evaluable lesions, including those that are not measurable
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
5. Adequately understand the study and voluntarily sign the Informed Consent Form;
6. ≥18 years old;
7. Lab tests within 7 days before first dose:

1) Absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥100×109/L, and hemoglobin ≥100g/L; 2) Serum total bilirubin ≤1.5 times the upper limit of normal (ULN); 3) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels ≤2.5 times the ULN； 4) Patients without anticoagulant therapy: International Normalized Ratio (INR) ≤1.5 ULN and activated partial thromboplastin time (APTT) ≤1.5 ULN. If patients received anticoagulant therapy: INR ≤2 ULN and APTT was within the normal range 14 days before treatment; 5) Serum total bilirubin <1.5 times the upper limit of normal (ULN); 6) Urine protein < 2+; if ≥2+, 24-hour urine protein <1 g; 8. Male or females patients with reproductive potential must agree to use an effective contraceptive method, for example, double-barrier device, condom, oral or injected birth control medication or intrauterine device, during the study and within 90 days after study treatment discontinuation. All female patients are considered to be fertile, unless the patient had natural menopause or artificial menopause or sterilization (such as hysterectomy, bilateral oophorectomy or ovarian irradiation).

Exclusion Criteria:

1. Prior system treatment with antiPD1/PDL1/PDL2/CTLA-4 antibody or Sulfatinib;
2. Previous intraperitoneal treatment with immunologic agents;
3. Patients with digestive tract obstruction or uncontrolled active bleeding from the primary tumor;
4. Patients with any active autoimmune disease or a documented history of autoimmune disease: Patients with hypothyroidism but receiving a stable dose of thyroid hormone replacement therapy were included in the study, and subjects with stable type 1 diabetes were able to control their blood sugar;
5. Pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-associated pneumonia, severe impaired lung function, etc;
6. Prior major surgery within past 4 weeks and had not fully recovered from previous surgery;
7. Active bleeding or abnormal coagulation, Prone to bleeding or receiving thrombolytic or anticoagulant therapy;
8. Hypertension that is not controlled by the drug, and is defined as: SBP≥140 mmHg and/or DBP≥90 mmHg;
9. Prior antitumor therapy (including chemotherapy, immunotherapy, biological treatment, Targeted therapy, etc) , or have not recovered from toxicities since the last treatment;
10. Pregnant or nursing;
11. previously received allogeneic stem cell or parenchymal organ transplantation;
12. Any significant clinical or laboratory abnormality that the investigator considers to influence the safety evaluators;
13. History of uncorrected serum electrolyte disturbances such as potassium, calcium, or magnesium;
14. Known human immunodeficiency virus (HIV) infection;
15. Active hepatitis B virus (HBV) and hepatitis C virus (HCV) infected persons;
16. A history of other malignancies within 5 years prior to inclusion, except for cervical carcinoma in situ, basal or squamous cell skin cancer, localized prostate cancer treated with radical surgery, and ductal carcinoma in situ treated with radical surgery;
17. Prior treatment with corticosteroids (dose > 10 mg/day prednisone or other hormones) or other immunosuppressive agents within 2 weeks, nasal or inhalation in allowed (dose > 10 mg/day prednisone or other hormones);
18. Severe, uncontrolled medical condition that would affect patients' compliance or obscure the interpretation of toxicity determination or adverse events, including active severe infection, uncontrolled diabetes, angiocardiopathy (heart failure > class II NYHA, LVEF <50%, myocardial infarction, unstable arrhythmia or unstable angina within past 6 months, cerebral infarction within past 3 months) or pulmonary disease ( interstitial pneumonia, obstructive pulmonary disease or symptomatic bronchospasm);
19. History with tuberculosis who are receiving or have received anti-TB treatment within 1 year;
20. Active infection;
21. Receiving another experimental drug or participating in a clinical study for another therapeutic purpose within the first 28 days prior to treatment initiation;
22. Any other disease, metabolic disorder, abnormal results of a physical examination or laboratory examination, and reasonably suspected disease or condition that may contraindication the use of the investigational drug, or affect the reliability of the study results, or place the patient at high risk for treatment complications, or affect patient compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of first dose of study drug until withdrawal of consent or death (up to approximately 1 year)
  Duration from the date of initial treatment with Surufatinib plus toripalimab to the date of death due to any cause.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anti-cancer therapy (up to approximately 1 year)
  A duration from the date of initial treatment with Surufatinib combined with Toripalimab to disease progression or death of any cause.
adverse events | 1 year
  Adverse events assessments are computed and categorized according to the Common Toxicity Criteria of the National Cancer Institute, version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No